CLINICAL TRIAL: NCT03674905
Title: Peripheral Nerve Block Compared to Intra-articular Injection for Post-operative Pain Control in Total Ankle Arthroplasty: A Randomized, Controlled Trial
Brief Title: Peripheral Nerve Block Compared to Intra-articular Injection for TAA Post-operative Pain
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Slocum Research & Education Foundation (Other)
Collaborators: Slocum Center for Orthopedics and Sports Medicine (Other)
Responsible Party: Principal Investigator, Nicholas Strasser, Principal Investigator, Slocum Research & Education Foundation
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: NLS_TAA1
Record Dates: First submitted 2018-09-11; First posted 2018-09-18 (Actual); Last update posted 2018-09-18 (Actual); Status verified 2018-09

CONDITIONS: Ankle Arthritis; Ankle Arthropathy
MeSH Terms: interventions — Injections, Intra-Articular

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Intra-articular injection (Other): Intra-articular injection at the completion of TAA procedure.
  Interventions: Procedure: Intra-articular injection
- Peripheral nerve block (Other): Pre-operative peripheral nerve block.
  Interventions: Procedure: Peripheral nerve block

INTERVENTIONS:
Procedure: Intra-articular injection — Intra-articular injection at the completion of TAA procedure.
  Arms: Intra-articular injection
Procedure: Peripheral nerve block — Pre-operative peripheral nerve block.
  Arms: Peripheral nerve block

SUMMARY:
Ankle arthritis is associated with debilitating pain and chronic disability. For the treatment of severe ankle arthritis, total ankle arthroplasty (TAA) is one treatment option. Postoperative pain management in joint arthroplasty is an ongoing and relevant issue. The purpose of this study is to examine if differences exist in postoperative pain control, overall patient satisfaction, and use of narcotics using an intra-articular injection in the operating room compared with a peripheral nerve block in patients undergoing TAA.

DETAILED DESCRIPTION:
This is a two-arm, prospective, randomized, controlled clinical study. Use of intra-articular injections in TAA are not widely reported in literature; however, they are commonly used during total knee arthroplasty's (TKAs). The purpose of this study is to examine if differences exist in postoperative pain control, overall patient satisfaction, and use of narcotics using the intra-articular injection compared with a peripheral nerve block in patients undergoing TAA. Results will contribute to the literature for the best surgical practice for pain management following a TAA for ankle arthritis.

Patients will be randomized to receive one of the following interventions for pain control in the operating room:

1. Intra-articular Injection
2. Preoperative Peripheral Nerve Block:

The study aims are:

* Aim 1: Determine if intra-articular injection as source of pain control for TAA lowers postoperative pain as measured by self-reported narcotic use and pain vs. the peripheral nerve block.
* Aim 2: Evaluate differences in functional outcomes and health related quality of life between intra-articular injections and peripheral nerve block as reported by pre- and post-operative patient questionnaires

Patients who consent to participate will complete study activities pre-operatively, and at 2 weeks, 6 weeks, and 3 months post-operatively.

ELIGIBILITY:
Inclusion Criteria:

* Patient is 40 - 80 years old
* Patient is having a primary, unilateral TAA
* Patient has signed the current, Institutional Review Board approved informed consent document

Exclusion Criteria:

* Patient has untreated endocrine disease
* Patient has uncontrolled diabetes; lab result of hemoglobin A1c level > 8.0 mg/dL
* Patient has significant heart, liver, kidney or respiratory disease
* Patient has peripheral vascular disease
* Patient has active cancer
* Patient has current history of narcotic use beyond that of oral medications
* Patient discharge status is known to be to care facility

Ages: 40 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 50 (Estimated)
Dates: Start 2016-11-29 (Actual); Primary Completion 2019-12 (Estimated); Study Completion 2020-12 (Estimated)

PRIMARY OUTCOMES:
Total narcotic use in morphine equivalents | Up to 3 months post-operatively
  Narcotic dose and frequency captured through patient diary; used to calculate morphine equivalents.
Self-reported pain captured with a visual analog pain scale | Up to 3 months post-operatively
  Measures self-reported pain between 0 (no pain) and 100 (extreme pain)

SECONDARY OUTCOMES:
Foot and Ankle Ability Measure (FAAM) | Up to 3 months post-operatively
  Measures self-reported outcomes accessing physical function for individuals with foot and ankle related impairments.
American Orthopaedic Foot and Ankle Society (AOFAS) Ankle Hindfoot Score | Up to 3 months post-operatively
  Grades ankle, subtalar, talonavicular, and calcaneocuboid joint levels in terms of pain (40 points), function (50 points), and alignment (10 points); 100 points possible sub-scores are summed, higher indicates better outcome.
Veterans Rand (VR) 36 item Health Survey | Up to 3 months post-operatively
  VR-36 Consists of select items from eight concepts of health in the VR-36, measuring health-related quality of life, and differences in disease burden.
Time to narcotic discontinuation | Up to 3 months post-operatively
  Number of days narcotics were taken for post-operative pain control

CONTACTS AND LOCATIONS:
Overall Officials: Nicholas L Strasser, MD, Principal Investigator — Slocum Center for Orthopedics and Sports Medicine
Locations (1):
- Slocum Research & Education Foundation, Eugene, Oregon, United States

IPD SHARING:
Plan to Share IPD: No